CLINICAL TRIAL: NCT04079010
Title: The Effect of Blood Flow Restriction With and Without Arginine on Physical Performance and Growth Hormone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mary Hardin-Baylor (Other)
Responsible Party: Principal Investigator, Kristi Trammell, Assistant Professor, Doctor of Physical Therapy program, University of Mary Hardin-Baylor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 57
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Blood Flow Restriction; Growth Hormone; Strength Outcomes; Arginine
Keywords: blood flow restriction; growth hormone; strength outcomes; arginine
MeSH Terms: interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Participants will adhere to resistance training protocol.
  Interventions: Dietary Supplement: Placebo Pill
- BFR (blood flow restriction) (Active Comparator): Participants will adhere to resistance training protocol, while also applying a blood flow restriction cuff during resistance training.
  Interventions: Procedure: BFR; Dietary Supplement: Placebo Pill
- BFR (blood flow restriction), plus Arginine (Active Comparator): Participants will adhere to resistance training protocol, apply a blood flow restriction cuff during resistance training, and will take the clinically safe dose of arginine prior to training sessions.
  Interventions: Procedure: BFR; Dietary Supplement: Arginine

INTERVENTIONS:
Procedure: BFR — Blood flow restriction (BFR) training is a non-invasive technique that uses wraps, bands, or inflated blood pressure cuffs to change blood flow within targeted muscles. Occlusion pressure of the femoral artery will be determine before each training session using the Delfi Personalize Tourniquet System for Blood Flow Restriction (2.0) which has embedded ultrasound technology to continually measure the blood flow and with auto-adjust the pressure. The target percent of occlusion is 50% of total blood flow while completed a prescribed resistance training regimen 4 times per week.
  Arms: BFR (blood flow restriction); BFR (blood flow restriction), plus Arginine
Dietary Supplement: Arginine — The BFR+Arg group will consume Arginine supplement daily throughout the course of the study. Supplements were manufactured by Kyowa, a US-based cGMP-compliant contract manufacturing facility independently audited and pre-qualified by the quality compliance firm, Obvium*Q, LLC (Dallas, TX). Manufacturing batch records for production of each of the supplements were maintained by the manufacturer and finished supplements were independently assayed for identity, purity, potency, and composition using appropriate USP, AOAC, or BAM methods at the independent, analytical laboratory, Dyad Labs (Salt Lake City, UT), prior to approval for release and consumption of the supplements by participants.
  Each serving of the supplements were formulated to contain 3,000 mg L-Arginine (ARG; Kyowa). Each supplement also contained the inert and non-insulinotropic excipient ingredients, microcystalline cellulose and silicon dioxide.
  Arms: BFR (blood flow restriction), plus Arginine
Dietary Supplement: Placebo Pill — The CON and BFR groups will consume placebo pill daily throughout the course of the study. Supplements were manufactured by Kyowa, a US-based cGMP-compliant contract manufacturing facility independently audited and pre-qualified by the quality compliance firm, Obvium*Q, LLC (Dallas, TX). Manufacturing batch records for production of each of the supplements were maintained by the manufacturer and finished supplements were independently assayed for identity, purity, potency, and composition using appropriate USP, AOAC, or BAM methods at the independent, analytical laboratory, Dyad Labs (Salt Lake City, UT), prior to approval for release and consumption of the supplements by participants.
  Each serving of the supplements were formulated to contain 3,000 mg Maltodextrin placebo (PLA; MALTRIN-M100; Grain Processing Corporation; Muscantine, IA). Each supplement also contained the inert and non-insulinotropic excipient ingredients, microcystalline cellulose and silicon dioxide.
  Other Names: Maltodextrose
  Arms: BFR (blood flow restriction); Control

SUMMARY:
The current study will investigate the effects of Blood Flow Restriction (BFR) training and L-arginine supplementation on recreationally trained female participants. In particular, it will compare performance outcomes and blood markers among two intervention groups (BFR and BFR+Arg) and a control group (CON).

DETAILED DESCRIPTION:
The current study will investigate the effects of Blood Flow Restriction (BFR) training and L-arginine supplementation on recreationally trained female participants. In particular, it will compare performance outcomes and blood markers among two intervention groups (BFR and BFR+Arg) and a control group (CON). All group will participate in the same training regimen. The control group will train and ingest a placebo pill. The BFR group will train with BFR and ingest a placebo pill, and the BFR+Arg group will train with BFR and ingest an L-arginine pill. All placebo pills will be Maltodextrin. The performance outcome is leg press 1RM, while the blood markers are growth hormone (GH) and cortisol. This analysis will provide insight as to whether or not L-arginine supplementation in addition to blood flow restriction training improves performance and muscle hypertrophy measure more than blood flow restriction training alone.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* PAR-Q form complete and without contraindications
* Body Mass Index (BMI) of 18.5-29.9 kg/m2
* Stable body weight prior to participation in the study (fluctuation not exceeding 10 lbs. within the past 6 months
* Agreement not to change current diet or exercise program (other than adding the program for the purpose of this study)

Exclusion Criteria:

* Any diagnosed orthopedic condition that prevents exercise
* BMI > 29.9 kg/m2 or < 18.5 kg/m2
* Affirmative answer to any of the questions presented on the PAR-Q form
* Are currently pregnant or planning to become pregnant during the study
* Currently taking blood pressure medication

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Strength | Baseline measurements will be obtained during Week 0, then measurements will be taken at Week 4 and Week 8 to determine the amount of change in participant's strength at those particular time points compared to baseline
  1 RM (rep-max) will be utilized to measure lower extremity strength

SECONDARY OUTCOMES:
Growth Factor | Measured at Week 0, Week 4, and Week 8 at the following intervals: prior to supplement, 15 and 30 minutes post-supplementation (before exercise), and 90 minutes post-supplementation (after exercise)
  Growth Hormone will be assessed by blood draw in an acute response design

OTHER OUTCOMES:
Cortisol | Measured at Week 0, Week 4, and Week 8 at the following intervals: prior to supplement, 15 and 30 minutes post-supplementation (before exercise), and 90 minutes post-supplementation (after exercise)
  Cortisol will be assessed by blood draw in an acute response design

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mary Hardin-Baylor, Belton, Texas, United States

IPD SHARING:
Plan to Share IPD: No